CLINICAL TRIAL: NCT05718167
Title: A Phase 3, Randomized, Double-blind, Parallel Controlled, Multi-center Study to Compare the Safety and Efficacy of TQB2450 Injection Combined With Paclitaxel Injection and Carboplatin Injection Followed by TQB2450 Injection Combined With Anlotinib Hydrochloride Capsules Versus Tislelizumab Injection Combined With Paclitaxel Injection and Carboplatin Injection Followed by Tislelizumab Injection as a First-line Treatment on Patient With Advanced Squamous NSCLC.
Brief Title: TQB2450 Injection Combined With Chemotherapy Followed by Sequential Combination With Anlotinib Hydrochloride Capsule for First-line Treatment of Advanced Squamous Non-small Cell Lung Cancer.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB2450-III-12
Record Dates: First submitted 2022-12-20; First posted 2023-02-08 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-04

CONDITIONS: Advanced Squamous Non-Small Cell Lung Carcinoma
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2450 Injection and Anlotinib Hydrochloride Capsules (Experimental): In the induction stage:
  TQB2450 injection: 1200 mg, Intravenous drip on d1; Carboplatin injection: Area Under Curve 5mg/mL/min, Intravenous drip on d1; Paclitaxel injection: 175mg/m2, Intravenous drip on d1. The above schemes are repeated every three weeks.
  In the maintenance stage:
  TQB2450 injection: 1200 mg, Intravenous drip on d1; Anlotinib Hydrochloride Capsules: 10mg, orally administered every day from d1-d14.
  The above schemes are repeated every three weeks.
  Interventions: Drug: TQB2450; Drug: Anlotinib hydrochloride capsule
- Tislelizumab Injection (Active Comparator): In the induction stage:
  Tislelizumab injection: 200 mg, Intravenous drip; Carboplatin injection: Area Under Curve 5mg/mL/min, Intravenous drip; Paclitaxel injection: 175mg/m2, Intravenous drip. The above schemes are repeated every three weeks.
  In the maintenance stage:
  Tislelizumab injection: 200 mg, Intravenous drip on d1 Placebo capsule: 0mg, orally administered every day from d1-d14. The above schemes are repeated every three weeks.
  Interventions: Drug: Tislelizumab injection

INTERVENTIONS:
Drug: TQB2450 — TQB2450 is a humanized monoclonal antibody targeting the programmed death ligand 1 (PD-L1), which prevents PD-L1 from binding to the PD-1 and B7.1 receptors on the surface of T cells, making T cells recover their activity, thereby enhancing the immune response.
  Arms: TQB2450 Injection and Anlotinib Hydrochloride Capsules
Drug: Anlotinib hydrochloride capsule — Anlotinib hydrochloride is a multi-target receptor tyrosine kinase inhibitor, which can target angiogenesis related kinases, such as VEGFR 1/2/3, FGFR 1/2/3 and other tumor cell proliferation related kinases like Platelet-derived growth factor receptor (PDGFR) α/β、 C-kit, RET.
  Arms: TQB2450 Injection and Anlotinib Hydrochloride Capsules
Drug: Tislelizumab injection — Tislelizumab injection can bind to human programmed cell death 1 (PD-1), a cell membrane protein that is mainly expressed on activated T cells and inhibits T cell activation.
  Arms: Tislelizumab Injection

SUMMARY:
This is Phase 3, randomized, double-blind, parallel controlled study designed to evaluate the Progression Free Survive (PFS) of TQB2450 injection combined with Paclitaxel Injection and Carboplatin Injection Followed by TQB2450 injection combined with Anlotinib Hydrochloride Capsules versus Tislelizumab injection combined with Paclitaxel Injection and Carboplatin Injection followed by Tislelizumab injection in locally advanced (stage ⅢB/ⅢC) and metastatic or recurrent (Stage IV) squamous NSCLC subjects.The primary endpoint is PFS assessed by IRC.

ELIGIBILITY:
Inclusion Criteria:

* According to the 8th edition of the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer Classification, the Tumour, node and metastasis (TNM) staging of lung cancer is locally advanced (stage ⅢB/ⅢC), metastatic or recurrent ( Stage IV) NSCLC patients.
* Between the ages of 18-75 years (calculated based on the date of signing ICF); male or female; Eastern cooperative oncology group (ECOG) score 0-1; estimated survival time ≥ 3 months.
* According to the RECIST 1.1 standard, there is at least one measurable lesion. If the measurable lesion is located in the radiotherapy area, it should be clearly defined as a progressive state.
* Patients who have not received systemic anti-tumor therapy for advanced, recurrent or metastatic diseases in the past. For those who have received adjuvant chemotherapy in the past, the interval between the recurrence time and the last adjuvant chemotherapy should be at least 6 months; The interval between the end of previous radiotherapy for chest and this treatment should be more than 6 months, and the interval between palliative radiotherapy for chest and this treatment should be more than 7 days.
* Tumor tissue sections that have not undergone radiotherapy at or after the diagnosis of advanced or metastatic NSCLC must be provided.These are Used for PD-L1 expression detection.Tumor tissue samples must be archived samples or freshly obtained samples within 12 months before randomization.
* main organ function is good, meet the following standards.

  1. Routine blood examination standards (without blood transfusion or correction with hematopoietic stimulating factor drugs within 14 days before screening):

     1. Absolute neutrophil count (ANC) ≥1.5×109 /L;
     2. Platelets ≥100×109 /L;
     3. Hemoglobin ≥90 g/L.
  2. The blood biochemical examination shall meet the following standards:

     1. Total bilirubin (TBIL) ≤ 2 × upper limit of normal (ULN) (Patients with Gilbert syndrome ≤ 3 × ULN);
     2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5×ULN. If it is accompanied by liver metastasis, ALT and AST≤5×ULN;
     3. Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance estimated by Cockcroft-Gault glomerular filtration formula ≥60 mL/min;
     4. Serum albumin (ALB) ≥30g/L.
  3. Urine routine examination standard: urine routine indicates urine protein <++; if urine protein ≥++, it is necessary to confirm that the 24-hour urine protein quantitative ≤1.0 g.
  4. Blood coagulation test standards: prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR)≤1.5×ULN (no anticoagulant therapy).
  5. Thyroid Stimulating Hormone (TSH) ≤ ULN; if abnormal, T3 and T4 levels should be examined. If T3 and T4 levels are normal, it can be selected.
  6. Heart color Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥50%.
  7. 12-lead ECG evaluation: QTc<450ms (male), QTc<470ms (female).
* Women of childbearing age should agree to use effective contraceptive measures during the study period and 6 months after the end of the study, and have a negative serum pregnancy test within 7 days before the study enrollment; men should agree to the study period and 6 months after the end of the study period Effective contraceptive measures must be used internally.
* The subjects voluntarily joined the study, signed the informed consent form, and had good compliance.

Exclusion Criteria:

* Tumor disease and medical history:

  1. Brain metastasis exists before enrollment. Subjects meeting one of the following requirements can be included;

     1. Have received brain metastasis treatment (surgery/radiotherapy) in the past and meet all the following criteria:

        * only supratentorial metastasis and cerebellar metastasis,
        * the condition needs to be stable for ≥ 2 weeks and no imaging evidence of new brain metastasis or brain metastasis expansion is found;
        * there is no brain metastasis symptom, and the subject must have stopped using corticosteroids/dehydrators for at least 2 weeks before starting to use the trial drug;
     2. The patient has not received brain metastasis treatment in the past and meets all the following criteria:

        * the maximum diameter of the lesion is less than 2cm;
        * the condition needs to be stable for ≥ 2 weeks (no imaging evidence of new brain metastasis or expanded brain metastasis is found), and there is no neurological symptoms caused by brain tissue compression;
        * the subject must have stopped using corticosteroids/dehydrating agents for at least 2 weeks before starting to use the test drug;
  2. There are midbrain, pons, medulla oblongata, spinal cord and meningeal metastases；
  3. Other malignant tumors appeared or were present within 3 years. The following two cases can be included: other malignant tumors treated by single operation have achieved 5-year Disease-free survival (DFS) in a row; The cured cervical carcinoma in situ, non melanoma skin cancer and superficial bladder tumor [ta (non-invasive tumor), tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
  4. Central type, cavity squamous cell carcinoma (primarily in the main bronchus and around the hilar);Imaging shows that the tumor invades large blood vessels or is unclearly separated from the blood vessels, or the investigator judges that the tumor is likely to invade important blood vessels and cause fatal bleeding during the subsequent study(The major vessels in the chest include pulmonary aorta, left pulmonary artery, right pulmonary artery, four pulmonary veins, superior vena cava, inferior vena cava and aorta);
  5. There is spinal cord compression and/or severe bone injury caused by tumor bone metastasis, including pathological fracture and severe bone pain with poor control;
  6. Patients with serous cavity (thoracic cavity, abdominal cavity, or pericardial cavity) that require repeated drainage to relieve clinical symptoms (as determined by the investigator), or who have received drainage of serous cavity effusion for the purpose of treatment within 2 weeks before treatment.
* Previous anti-tumor treatments:

  1. Received the treatment of proprietary Chinese medicines with anti-tumor indications specified in the China National Medical Products Administration (NMPA) approved drug instructions within 2 weeks before the start of the study treatment(Including compound cantharidin capsules, Kangai injection, Kanglaite capsule/injection, Aidi injection, brucea javanica oil injection/capsule, Xiaoaiping tablet/injection, Huachansu capsule, etc.);
  2. Previously received related immunotherapy drugs for programmed death 1 (PD-1), PD-L1, cytolytic T lymphocyte-associated antigen-4 (CTLA-4), etc.;
  3. Previous use of anti-angiogenic drugs such as bevacizumab, anlotinib, apatinib, lenvatinib, sorafenib, sunitinib, regorafenib, fruquintinib, etc.;
  4. Failure to recover from the toxicity and/or complications of previous interventions to CTCAE ≤1, except for hair loss and peripheral neuropathy ≤2;
* Combined diseases and medical history:

  1. Liver cirrhosis, active hepatitis*;(Note: active hepatitis (hepatitis B reference: HBV-DNA > 1*103 copy /mL or > 2000IU/mL) when HBsAg is positive. Hepatitis C reference: Hepatitis C virus (HCV) antibody is positive, and HCV titer detection value exceeds the upper limit of normal value);
  2. Renal abnormalities: i.Renal failure requires hemodialysis or peritoneal dialysis; ii.Previous or existing nephrotic syndrome, chronic nephritis.
  3. Cardiovascular and cerebrovascular abnormalities：

     1. Patients with previous or present heart failure, degree II or above heart block:
     2. Myocardial infarction or unstable angina, supraventricular or ventricular arrhythmia with clinical significance need treatment or intervention;
     3. Vascular embolism and cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage and cerebral infarction) occurred within 9 months（ Prophylactic use of anticoagulant therapy is allowed for patients with thrombotic tendency or undergoing anticoagulant therapy.)
     4. After more than two kinds of drug treatment, blood pressure control is still not ideal (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 90 mmHg).
  4. Gastrointestinal abnormalities:

     1. Inability to take medications (such as inability to swallow, intestinal obstruction, etc.);
     2. A history of malabsorption syndrome or other diseases that interfere with gastrointestinal absorption;
     3. Received treatment for active peptic ulcer in the past 6 months;
     4. Despite the maximum medical treatment, chronic diarrhea of grade 2 and above continues to occur;
     5. Other conditions determined by the researcher that may cause gastrointestinal bleeding and perforation.
  5. History of immunodeficiency:

     1. Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases;
     2. Active autoimmune disease or history of autoimmune disease, including but not limited to Crohn's disease, ulcerative colitis, autoimmune hepatitis/enteritis/vasculitis/nephritis, etc.
     3. Prepare to undergo or have previously received an organ transplant;
     4. Patients who require systemic or topical immunosuppressive therapy to achieve immunosuppressive purposes and need to continue to use them within two weeks before randomization (except for glucocorticoid daily dose <10 mg prednisone or other equivalent hormones). (Note: Hormone replacement therapy (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered as systemic therapy and allowed to be used.)
  6. Bleeding risk:

     1. Suffered from bleeding or coagulopathy within 28 days before the start of treatment or was using warfarin, aspirin and other antiplatelet agglutination drugs (except for aspirin ≤100 mg/d preventive drugs);
     2. Had hemoptysis >2.5 mL/day in 28 days before the start of treatment;
     3. Regardless of the severity, patients with any history of bleeding or coagulopathy;
     4. Received major surgical treatment, open biopsy, etc. within 28 days before the start of the study treatment;
     5. Long-term unhealed wounds or fractures, except for pathological fractures;
  7. Poor control of type I diabetes or II diabetes (fasting blood glucose (FBG)> 10mmol/L);
  8. Severe infections within 4 weeks before the start of study treatment, including but not limited to hospitalization due to bacteremia, severe pneumonia, or other severe infections; subjects with ≥ grade 2 active infections within 4 weeks before the start of study treatment Or fever of unknown cause occurred during the screening period and before the first administration>38.0℃;
  9. Past or existing pneumoconiosis, interstitial pneumonia, (non-infectious) pneumonia that requires adrenal corticosteroid therapy, currently suffering from other types of pneumonia ≥2, or lung function tests confirmed severely impaired lung function (Forced Expiratory Volume in the first second (FEV1) or diffusing capacity of lung for carbon monoxide(DLCO) or DLCO per alveolar volume (DLCO /VA) accounts for the expected value %<40%) and other objective evidence;
  10. Patients with active tuberculosis within 1 year before enrollment; subjects with a history of active pulmonary tuberculosis infection 1 year ago must provide clear evidence of cure before enrollment; if tuberculosis is suspected during the screening period, chest radiographs and sputum must be passed Enter the group only after the liquid and clinical symptoms are eliminated;
  11. Allergies, or a history of severe allergies in the past, or severe hypersensitivity reactions after receiving other monoclonal antibody treatments, or known allergies to the ingredients of the study drug excipients;
  12. Previous history of severe mental disorders;
  13. People with a history of drug abuse, alcohol or drug abuse;
* The end of the previous clinical study (last dose) is less than 4 weeks or the study drug's 5 half-lives, whichever is shorter.
* Live attenuated vaccine vaccination history within 28 days before randomization or planned live attenuated vaccination during the study period. Seasonal influenza vaccine for injection is usually an inactivated virus vaccine and is allowed to be vaccinated during the study period.
* Female patients during pregnancy or lactation.
* For patients with known epidermal growth factor receptor (EGFR) sensitive mutation, anaplastic lymphoma kinase (ALK) fusion and ROS proto-oncogene 1 (ROS1) fusion, detection is not mandatory for those with unknown gene status
* According to the investigator's point of view, it may increase the risks associated with participating in the study, or other severe, acute or chronic medical diseases or laboratory abnormalities that may interfere with the interpretation of the study results, or other reasons that are not suitable for participating in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Base line up to 2 years. The curative effect was evaluated every 6 weeks (42 days) in the first 54 weeks of treatment period; After 54 weeks, the efficacy was evaluated every 9 weeks (63 days).
  Progression Free Survival (PFS) assessed by Independent Review Committee (IRC)

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline up to death event, assessed up to 2 years.
  Overall survival is the time from randomization to the time of death from any cause.
Progression free survival (PFS) | From randomization to Progression disease, assessed up to 2 years.
  Progression free survival (PFS) assessed by investigators according to The Response Evaluation Criteria In Solid Tumors 1.1 (RECIST) and iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics.
Objective response rate (ORR) | From randomization to Progression disease, assessed up to 2 years.
  Objective response rate (ORR), assessed by investigators according to The Response Evaluation Criteria In Solid Tumors 1.1 (RECIST) and iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics.
Disease control rate (DCR) | From randomization to Progression disease, assessed up to 2 years.
  Disease control rate (DCR)assessed by investigators according to RECIST 1.1 and iRECIST criteria
Duration of response (DOR) | From randomization to Progression disease, assessed up to 2 years.
  Duration of response (DOR) assessed by investigators according to RECIST1.1 and iRECIST criteria
The occurrence of all adverse events (AEs) | Baseline up to 2 years.
  The occurrence of adverse events (AEs) is to evaluate safety profile
The severity of all adverse events (AEs) | Baseline up to 2 years.
  The severity of adverse events (AEs) is to evaluate safety profile
The occurrence of abnormal heart rate in 12 lead Electrocardiograph (ECG) | Baseline up to 2 years.
  The occurence of abnormal heart rate is to evaluate safety profile
The severity of abnormal heart rate in 12 lead Electrocardiograph (ECG) | Baseline up to 2 years.
  The severity of abnormal heart rate is evaluated in accordance with the standard of common toxic reactions of the National Cancer Institute [NCI CTC v5.0].
The occurrence of abnormal PR interval in 12 lead ECG | Baseline up to 2 years.
  The occurrence rate of abnormal 12 lead ECG is to evaluate safety profile. The results of PR interval were divided into low, normal and high according to the normal value range.
The severity of abnormal PR interval in 12 lead ECG | Baseline up to 2 years.
  The results of PR interval were divided into low, normal and high according to the normal value range, and the relative baseline change was described with a cross table. The minimum or maximum observed value after the baseline is used to calculate the results after the baseline.
  Descriptively summarize the results of PR examination at each visit, classify them as normal, abnormal without clinical significance, and abnormal with clinical significance, and compare them with the results of baseline, and describe them with cross classification table. The severity is evaluated in accordance with the standard of common toxic reactions of the National Cancer Institute [NCI CTC v5.0]
The occurrence of abnormal QRS interval in 12 lead ECG | Baseline up to 2 years.
  The occurrence of abnormal 12 lead ECG is to evaluate safety profile. The QRS interval results were divided into low, normal and high according to the normal value range.
The severity of abnormal QRS interval in 12 lead ECG | Baseline up to 2 years.
  The QRS interval results were divided into low, normal and high according to the normal value range, and the relative baseline change was described with a cross table. The minimum or maximum observed value after the baseline is used to calculate the results after the baseline.
  Descriptively summarize the results of PR examination at each visit, classify them as normal, abnormal without clinical significance, and abnormal with clinical significance, and compare them with the results of baseline, and describe them with cross classification table. The severity is evaluated in accordance with the standard of common toxic reactions of the National Cancer Institute [NCI CTC v5.0]
The occurrence of abnormal QT interval in 12 lead ECG | Baseline up to 2 years.
  The occurrence rate of Abnormal 12 lead ECG is to evaluate safety profile. The results of QT interval were divided into low, normal and high according to the normal value.
The severity of abnormal QT interval in 12 lead ECG | Baseline up to 2 years.
  The results of QT interval were divided into low, normal and high according to the normal value range, and the relative baseline change was described with a cross table. The minimum or maximum observed value after the baseline is used to calculate the results after the baseline.
  Descriptively summarize the results of PR examination at each visit, classify them as normal, abnormal without clinical significance, and abnormal with clinical significance, and compare them with the results of baseline, and describe them with cross classification table. The severity is evaluated in accordance with the standard of common toxic reactions of the National Cancer Institute [NCI CTC v5.0]
The occurrence of abnormal QTc interval in 12 lead ECG | Baseline up to 2 years.
  The occurrence of Abnormal 12 lead ECG is to evaluate safety profile. The results of QTc interval were divided into low, normal and high according to the normal value.
The severity of abnormal QTc interval in 12 lead ECG | Baseline up to 2 years.
  The results of QTc interval were divided into low, normal and high according to the normal value range, and the relative baseline change was described with a cross table. The minimum or maximum observed value after the baseline is used to calculate the results after the baseline.
  Descriptively summarize the results of PR examination at each visit, classify them as normal, abnormal without clinical significance, and abnormal with clinical significance, and compare them with the results of baseline, and describe them with cross classification table. The severity is evaluated in accordance with the standard of common toxic reactions of the National Cancer Institute [NCI CTC v5.0]
The occurrence of serious adverse events (SAEs) | Baseline up to 2 years.
  The occurrence of serious adverse events (SAEs) is to evaluate safety profile
The severity of serious adverse events (SAEs) | Baseline up to 2 years.
  The severity of serious adverse events (SAEs) is to evaluate safety profile
European organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ-C30) | Baseline up to 2 years.
  QLQ-C30 is a quality of life questionnaire to help understand the physical condition of the subjects. The subjects need to answer them in person and circle the number that best reflects their situation. Among them, 1 represents no, 2 represents a little, 3 represents some, and 4 represents a lot. Questions 29 and 30 need to choose the most suitable number from 1 to 7 and draw a circle. The other 1 represents very poor, and 7 represents very good. Questions 29 and 30 need to choose the most suitable number from 1 to 7 and draw a circle. The other 1 represents very poor, and 7 represents very good.
Quality of life questionnaire lung cancer module (QLQ-LC13) | Baseline up to 2 years.
  QLQ-LC13 is a quality of life questionnaire to help understand the physical condition of the subjects. The subjects need to answer them in person and circle the number that best reflects their situation. Among them, 1 represents no, 2 represents a little, 3 represents some, and 4 represents a lot.
EuroQol Five Dimensions Questionnaire (EQ-5D) assessment pro | Baseline up to 2 years.
  EQ-5D assessment pro is a quality of life questionnaire, which has five questions that need to be answered by the subjects themselves, choose the answer that best reflects their health, and mark the point on the set scale that best represents their health, of which 100 represents the best condition and 0 represents the worst condition.
Incidence of Antidrug antibody | Baseline up to 2 years.
  It's a parameter to evaluate the immunogenicity of TQB2450 injection
Incidence of neutralizing antibody | Baseline up to 2 years.
  It's a parameter to evaluate the immunogenicity of TQB2450 injection

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - TianJin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan